CLINICAL TRIAL: NCT04874168
Title: The Efficacy of Transversus Abdominis Plane Block Versus Wound Infiltration for Analgesia After Cesarean Delivery: (A Randomized Controlled Double-blinded Clinical Trial )
Brief Title: The Efficacy of Transversus Abdominis Plane Block Versus Wound Infiltration for Analgesia After Cesarean Delivery:
Acronym: TAPBLOCK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Mohamed Mostafa, Clinical professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tapblockvwoundInfiltration
Record Dates: First submitted 2021-04-25; First posted 2021-05-05 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: computer-generated table of random numbers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In the TAP group (Group A ) (Active Comparator): after completion of surgery, bilateral ultrasound-guided TAP block was performed .
  Description of the intervention: a 12-4-MHz linear array transducer (ClearVue 350; Philips, Bothell, WA) placed transversely between the iliac crest and costal margin in the anterior axillary line and slid medial-lateral to visualize the external oblique, internal oblique, and trans-versus abdominis muscles; the most lateral (posterior) position obtaining a satisfactory ultrasound image was used ;A 22-gauge spinal needle was introduced from medial to lateral in-plane to the ultrasound probe, and 20 mL of bupivacaine 0.25% was injected under visualization in the plane between the transversus abdominis muscle and the fascia deep to the internal oblique muscle on each side.
  Interventions: Device: TAP block
- In the infiltration group (Group B ) (Active Comparator): at the end of surgery, 40 mL of bupivacaine 0.25% was injected subcutaneously in the surgical wound (20 mL in each of the upper and lower sides) by the obstetrician before skin closure.
  Interventions: Device: TAP block
- In placebo group (Group C ) (Placebo Comparator): routine analgesic was administered and recorded .
  Interventions: Device: TAP block

INTERVENTIONS:
Device: TAP block — bilateral ultrasound-guided TAP block was performed using a 12-4-MHz linear array transducer (ClearVue 350; Philips, Bothell, WA) placed transversely between the iliac crest and costal margin in the anterior axillary line and slid medial-lateral to visualize the external oblique, internal oblique, and trans-versus abdominis muscles; the most lateral (posterior) position obtaining a satisfactory ultrasound image was used
  Other Names: wound infiltration

SUMMARY:
This study aimed to compare bilateral ultrasound-guided TAP block with single-shot local anesthetic wound infiltration for analgesia after cesarean delivery performed under spinal anesthesia

DETAILED DESCRIPTION:
This double-blind, randomized controlled trial aimed to compare bilateral ultrasound-guided TAP block to single-shot local anesthetic wound infiltration for analgesia after cesarean delivery performed under spinal anesthesia. This will be done by measuring VAS (visual analogue score) for pain after ceserian section at2, 4, 6, 12, 24 hours .

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing cesarean section under spinal anesthesia
* Aged ≥19 years and > 40 years .
* Gestational age ≥ 37 Weeks .
* Informed Consent From the Patient .

Exclusion Criteria:

* Body mass index (BMI) ≥40 kg/m2 ..
* History of recent opioid exposure .
* Hypersensitivity to any of the drugs used in the study .
* Significant cardiovascular, renal, or hepatic disease.

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing cesarean section under spinal anesthesia .
Enrollment: 210 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The degree of pain at rest ; | From 2 hours to 24 hours postoperatively
  using an Visual analogue scale (VAS) scores for pain intensity reported on 0-10 point scale for analysis. (0 = no pain and 10 = the worst possible pain) .

SECONDARY OUTCOMES:
The time to the first postoperative opioid dose | at 2, 4, 6, and 12 hours.
  cumulative opioid consumption

OTHER OUTCOMES:
The degree of pain on movement (hip flexion and coughing) | From 2 hours to 24 hours postoperatively
  using an Visual analogue scale (VAS) scores for pain intensity reported on 0-10 point scale for analysis. (0 = no pain and 10 = the worst possible pain) .

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed G Elnajar, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Alabbasia, Egypt

IPD SHARING:
Plan to Share IPD: No